CLINICAL TRIAL: NCT05583617
Title: A Platform Study Evaluating the Safety and Efficacy of Multiple Treatments in Patients With Multiple Myeloma
Brief Title: A Study Evaluating the Safety and Efficacy of Multiple Treatments in Participants With Multiple Myeloma
Acronym: PLYCOM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CO43923; 2021-005918-34 (EudraCT Number); 2023-504484-16-00 (EU CTIS Number)
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; tocilizumab; iberdomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Substudy 2: Dose Escalation and Expansion (Experimental): In the pre-phase, participants will receive 2 step-up doses and a target dose of cevostamab. The step-up dose will be given on Day(D)1 and D4. The target dose will be given on D8. Subsequently the target dose will be administered on D1 and D15 for cycles 1-6 and D1 of cycle 7 onwards. Each cycle is 28 days. Lenalidomide will be administered by mouth (PO) on a 28-day cycle.
  During the dose expansion phase, cevostamab will be administered following the same dosing schedule as the dose escalation phase. The target dose will be determined after the escalation phase. Lenalidomide will be administered PO on a 28-day cycle.
  Enrollment for Substudy 2 has closed.
  Interventions: Drug: Cevostamab; Drug: Lenalidomide; Drug: Tocilizumab
- Substudy 4: Dose Escalation and Expansion (Experimental): In the pre-phase, participants will receive 2 step-up doses and a target dose of cevostamab. The step-up dose will be given on D1 and D4. The target dose will be given on D8. Subsequently the target dose will be administered on D1 of each cycle, every 3 weeks (Q3W). Each cycle is 21 days. Iberdomide will be administered PO on a 21-day cycle.
  During the dose expansion phase, cevostamab will be administered following the same dosing schedule as the dose escalation phase. The target dose will be determined after the escalation phase. Iberdomide will be administered PO on a 21-day cycle.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab; Drug: Iberdomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cevostamab — Substudy 2: Cevostamab will be administered intravenously (IV) on a 28-day cycle, up to a total of 13 cycles.
  Substudy 4: Cevostamab will be administered by IV on a 21-day cycle, up to a total of 17 cycles.
Drug: Lenalidomide — Lenalidomide will be administered PO on days 1-21 of a 28-day cycle.
  Arms: Substudy 2: Dose Escalation and Expansion
Drug: Tocilizumab — Tocilizumab will be administered for the treatment of cytokine release syndrome (CRS) when necessary.
Drug: Iberdomide — Iberdomide will be administered PO on days 1-14 of a 21-day cycle.
  Arms: Substudy 4: Dose Escalation and Expansion
Drug: Dexamethasone — Dexamethasone will be administered on Days 2 and 8 of Cycles 1-3.
  Arms: Substudy 4: Dose Escalation and Expansion

SUMMARY:
CO43923 is a platform study that will evaluate the safety, efficacy, and pharmacokinetics (PK) of multiple treatment combinations, as monotherapy or in combination, in participants with multiple myeloma (MM). The study is designed with the flexibility to open new treatment substudies as new treatments become available. Information regarding the opened substudies are found below.

DETAILED DESCRIPTION:
Cevos + Len substudy(SS) 2 (DIRAC):

This substudy will explore the combination of cevostamab and lenalidomide as post-transplant maintenance therapy in participants with MM with high-risk cytogenetic features who experienced at least a partial response (PR) after induction.

Cevostamab + Iberdomide SS4 (CHAWLA):

This substudy will evaluate the safety, tolerability, PK, and pharmacodynamics of the combination of cevostamab and iberdomide in participants with R/R MM who have received at least three prior lines of therapy, including a PI, an IMiD, and an anti-CD38 monoclonal antibody.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MM per International Myeloma Working Group (IMWG) criteria
* Eastern Cooperative Oncology Group Performance Status of 0, or 1, or 2
* Resolution of AEs from prior anti-cancer therapy to Grade <=1
* Agreement to undergo scheduled assessments and procedures

Additional Inclusion Criteria for SS2:

* Completion of planned induction therapy and achievement of at least a partial response (PR)
* Autologous Stem Cell Transplant (SCT) within 100 days prior to first study treatment and the absence of progressive disease
* Cytogenetic high-risk features at diagnosis
* Treatment with any investigational medicinal products, systemic cancer therapies, immunotherapies received previously in CO43923 (any arms) within 5 half-lives or 3 weeks whichever is the shortest
* Agreement to comply with all local requirements of the lenalidomide risk minimization plan, which includes the global pregnancy prevention program
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom even if they have had a prior vasectomy, and agreement to refrain from donating sperm

Additional Inclusion Criteria for SS4:

* Previously exposed to at least a PI, an IMiD, and an anti-CD38 antibody for the treatment of R/R MM for whom no suitable SOC therapy options are available

Exclusion Criteria:

* Inability to comply with protocol-mandated hospitalization and procedures
* History of confirmed progressive multifocal leukoencephalopathy
* History of other malignancy within 2 years prior to screening
* Current or past history of central nervous system (CNS) disease
* Significant cardiovascular disease that may limit a participant's ability to adequately respond to a CRS event
* Symptomatic active pulmonary disease or requiring supplemental oxygen
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection at study enrollment, or any major episode of infection requiring treatment with IV antibiotics where the last dose of IV antibiotics was given within 14 days prior to first study treatment
* Known or suspected chronic active Epstein-Barr virus (EBV) infection
* Positive serologic or PCR test results for acute or chronic hepatitis B virus (HBV) infection
* Acute or chronic hepatitis C virus (HCV) infection
* Known history of HIV seropositivity
* Administration of a live, attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipation that such a live, attenuated vaccine will be required during the study
* Any medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Additional Exclusion Criteria for SS2:

* Hypersensitivity reactions to lenalidomide or other immunomodulatory drugs
* Harbor lesions at proximity of vital organs that may develop sudden decompensation/deterioration in the setting of a tumor flare
* Prior treatment with any investigational medicinal product, systemic cancer therapy, or immunotherapies in any arm of study CO43923 within 5 half-lives or 3 weeks, whichever is shorter
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antimicrobials where the last dose of IV antimicrobial was given within 14 days prior to first study treatment
* History of erythema multiforme, Grade >=3 rash, or blistering following prior treatment with immunomodulatory derivatives
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the final dose of study treatment Exlcusion Criteria Applicable to SS2 and SS4
* History of autoimmune disease
* Known history of hemophagocytic lymphohistiocytosis (HLH) or macrophage activation syndrome (MAS)
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Received a cumulative dose of corticosteroids equivalent to >=140 mg of prednisone within the 14-day period before the first dose of the study drug (does not include pretreatment medication)
* Active symptomatic COVID-19 infection at study enrollment or requiring treatment with IV antiviral where the last dose of IV antiviral treatment was given within 14 days prior to first study treatment. Participants with active COVID-19 infection must have clinical recovery and two negative antigen tests at least 24 hours apart prior to first study treatment.
* Positive and quantifiable EBV PCR or CMV PCR prior to first study treatment

Additional Exclusion Criteria for SS4:

* Treatment with any investigational medicinal products, systemic cancer therapies, immunotherapies within 5 half-lives or 12 weeks before starting pre-phase
* History of anaphylaxis or hypersensitivity, including >=Grade 3 rash, during prior treatment with IMiDs, dexamethasone, any CELMoDs, or the excipients contained in the formulations
* Known anaphylaxis, allergies, hypersensitivity, or intolerance to boron or mannitol, hyaluronidase, sorbitol, corticosteroids, monoclonal antibodies (or recombinant antibody-related fusion proteins), or human proteins, CRBN modulating agents or their excipients, or known sensitivity to mammalian-derived products
* Administration of strong CYP3A modulators; administration of proton-pump inhibitors within 2 weeks of starting study treatment
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment
* Concurrent administration of a strong inhibitor, modulator or inducer of cytochrome P450 (CYP3A4/5) (including within 14 days of initiating study treatment)
* History of malignancies, other than MM, unless the subject has been free of the disease for >=5 years
* Peripheral neuropathy >Grade 2
* Prior treatment with cevostamab or another agent targeting FcRH5 or iberdomide
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the final dose of study treatment
* History of Stevens-Johnson syndrome, toxic epidermal necrolysis, or drug rash with eosinophilia and systemic symptoms
* Treatment with systemic immunosuppressive medications
* Prior treatment with CAR T-cell therapy (autologous or allogeneic) within 12 weeks before starting pre-phase
* Autologous SCT within 100 days prior to starting pre-phase
* Prior allogeneic SCT
* Plasmacytoma in proximity of vital organs that may develop sudden decompensation/deterioration in the setting of a tumor flare

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Percentage of Participants with Adverse Events (AEs) | Baseline up to approximately 5 years
Stage 2: Objective Response Rate (ORR) | Baseline up to approximately 5 years
Stage 2: Complete Response (CR) or Stringent Complete Response (sCR) Rate | Baseline up to approximately 5 years
Stage 2: Rate of Very Good Partial Response (VGPR) or Better | Baseline up to approximately 5 years
Stage 2: Progression-free Survival (PFS) | Baseline up to approximately 5 years
Stage 2: Overall Survival (OS) | Baseline up to approximately 5 years

SECONDARY OUTCOMES:
Stage 1: Conversion to a Better Response | Baseline up to approximately 5 years
Stage 1: PFS | Baseline up to approximately 5 years
Stages 1 and 2: Duration of Response (DOR) | Baseline up to approximately 5 years
Stage 1: OS | Baseline up to approximately 5 years
Stages 1 and 2: Minimal Residual Disease (MRD) Negativity Rate | Baseline up to approximately 5 years
Stage 1: ORR | Baseline up to approximately 5 years
Stage 1: CR or sCR Rate | Baseline up to approximately 5 years
Stage 1: Rate of VGPR or Better | Baseline up to approximately 5 years
Stage 2: Stage 1: Percentage of Participants with AEs | Baseline up to approximately 5 years
Stages 1 and 2: Time to First Response (for Participants who Achieve a Response of PR or Better) | Baseline up to approximately 5 years
Stages 1 and 2: Time to Best Response (for Participants who Achieve a Response of PR or Better) | Baseline up to approximately 5 years
Stages 1 and 2: Maximum Concentration Observed (Cmax) | Baseline up to approximately 5 years
Stages 1 and 2: Minimum Concentration under Steady-State Conditions within a Dosing Interval (Cmin) | Baseline up to approximately 5 years
Stages 1 and 2: Time to Maximum Concentration (Tmax) | Baseline up to approximately 5 years
Stages 1 and 2: Area under the Concentration-Time Curve (AUC) | Baseline up to approximately 5 years
Stages 1 and 2: Total Clearance of Drug (CL) | Baseline up to approximately 5 years
Stages 1 and 2: Volume of Distribution at Steady State | Baseline up to approximately 5 years
Stages 1 and 2: Terminal half-life | Baseline up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- Australia (2):
  - Prince of Wales Hospital, Randwick, New South Wales
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- France (4):
  - CHU Lyon Sud - Service Hématologie, Pierre-Bénite
  - IUCT Oncopole, Toulouse
  - Hopital Bretonneau, Tours
  - IGR, Villejuif
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf Onkologisches Zentrum Medizinische Klinik II, Hamburg
  - Universitätsklinikum Leipzig - Klinik und Poliklinik für Hämatologie, Leipzig
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Oddzial Kliniczny Hematologii SPZOZ MSWiA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Późna
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing